CLINICAL TRIAL: NCT03262519
Title: The Effect of Obstructive Sleep Apnea and Its Treatment on Decision Making
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Assistant Clinical Professor, University of California, San Diego
Other Study IDs: 170683
Record Dates: First submitted 2017-07-25; First posted 2017-08-25 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients at UCSD Sleep Medicine Clinic: Patients referred for sleep testing (either home sleep testing or in-lab full polysomnography) will be approached for participation.
  Interventions: Diagnostic Test: Computer based neurocognitive testing

INTERVENTIONS:
Diagnostic Test: Computer based neurocognitive testing — Iowa Gambling Task, The Balloon Task, Intertemporal choices task, Cognitive Reflection Test, Physiological and self-reported measures of OSA/sleep related symptoms, General health and physiological measures.

SUMMARY:
Obstructive sleep apnea (OSA) is an extremely common disease with inadequately explored neurocognitive consequences. The investigators will study OSA patients before and after treatment to understand how OSA changes decision making abilities, and whether treatment can reverse such cognitive changes. These results could provide deeper insight into how OSA affects decision making either temporarily or permanently, and provide another rationale or motivation for treatment of OSA in adults.

DETAILED DESCRIPTION:
The investigators hypothesize that OSA will lead to (H1) more reward-seeking and lower payoffs in the Iowa Gambling task, replicating previous findings; (H2) greater discounting of future rewards in financial choices; and (H3) these effects would dissipate when OSA is successfully treated.

In order to test these hypotheses, the investigators will perform cognitive tests (Iowa gambling; intertemporal choice; other measures) in 100 patients about to undergo sleep testing. It is expected that of these 100 patients, some will have no sleep apnea; some will have sleep apnea and will be successfully treated; and that some will have sleep apnea but will not be successfully treated by the time of repeat testing. The investigators will repeat testing using the same instruments 2 months later.

Thus the investigators will be able to compare whether OSA patients differ from control at baseline (t1), and whether OSA patients' performance will improve after treatment at t2, compared to the control at t2.

ELIGIBILITY:
Inclusion Criteria:

Subjects aged 18-75 referred to the UCSD Sleep clinic for either home or in-laboratory testing will be considered for inclusion in the study. Inclusion will not depend on gender, race or ethnicity, as per the following:

1. 100 participants will be enrolled at the UCSD Sleep Clinic at Chancellor Park.
2. Ages 18-75
3. Gender: Men and woman
4. Ethnic background: All
5. Health Status: to the UCSD Sleep clinic for either home or in-laboratory testing

Exclusion Criteria:

1. Ongoing CPAP treatment for OSA
2. Inability to use a tablet device (e.g. no reading glasses, or unfamiliar with devices).
3. Severe cardiopulmonary disorder that requires treatment with supplemental oxygen therapy.
4. Inability to speak English fluently, as some of the questionnaires/tests are only validated in English.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged 18-75 referred to the UCSD Sleep clinic for either home or in-laboratory testing will be considered for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Iowa Gambling Task | 2 months (baseline, 2 months later)
  The Iowa Gambling Task is a psychological task thought to simulate real-life decision making. It is completed on a computer and takes about 10 minutes. It is widely used in research on cognition.

SECONDARY OUTCOMES:
Change in Cognitive Reflection Test (CRT) | 2 months (baseline, 2 months later)
  The Cognitive Reflection Test (CRT) is a task designed to measure a person's tendency to override an incorrect "gut" response and engage in further reflection to find a correct answer. It takes about 3 minutes to complete.
Change in Intertemporal Choice | 2 months (baseline, 2 months later)
  Intertemporal choice is the study of how people make choices about what and how much to do at various points in time, when choices at one time influence the possibilities available at other points in time. These choices are influenced by the relative value people assign to two or more payoffs at different points in time. It takes about 3 minutes to complete.
Change in Balloon Analogue Risk Task (BART) | 2 months (baseline, 2 months later)
  The Balloon Analogue Risk Task (BART) is a computerized measure of risk taking behavior. The BART models real-world risk behavior through the conceptual frame of balancing the potential for reward versus loss. It takes less than 2 minute to complete.
Change in Epworth Sleepiness Score | 2 months (baseline, 2 months later)
  An 11 item questionnaire that is commonly used to assess for excessive daytime sleepiness (range 0-24 points, >10 considered excessively sleepy).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided